CLINICAL TRIAL: NCT03304405
Title: Influence of Sagittal Imbalance of the Spine on Gait Pattern in Adult Spinal Deformity
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Kenny Kwan, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW 16-294
Record Dates: First submitted 2017-09-27; First posted 2017-10-09 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Adult Spinal Deformity
Keywords: ASD
MeSH Terms: interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gait Analysis: All patients will undergo gait analysis using reflective surface markers placed at different locations on the head, trunk, upper and lower extremities, and pelvis. All patients will complete an analog pain scale, Oswestry, and SRS-22 questionnaires. These are health-related quality of life questionnaires that provide subjective assessment.
  Interventions: Diagnostic Test: Gait Analysis

INTERVENTIONS:
Diagnostic Test: Gait Analysis — All patients will undergo gait analysis using reflective surface markers placed at different locations on the head, trunk, upper and lower extremities, and pelvis. All patients will complete an analog pain scale, Oswestry, and SRS-22 questionnaires. These are health-related quality of life questionnaires that provide subjective assessment.

SUMMARY:
This study intends to investigate the changes in gait pattern in adult spinal deformity (ASD) patients with sagittal imbalance. It will investigate the gait kinematics in patients who have a mismatch of their spinopelvic parameters, and a positive sagittal balance. The investigators hypothesise that patients with abnormal spinopelvic parameters may demonstrate a pathological gait pattern.

DETAILED DESCRIPTION:
With an ageing population, ASD presents as a significant health issue with increasing incidence. Most of the earlier literature concentrated on radiographic measurements of the deformity in the coronal plane, and its surgical correction. However, recent publications have demonstrated that sagittal spinopelvic alignment plays a critical role in pain and disability in patients with ASD, and is a primary determinant of health related quality of life measures. There is substantial evidence that restoration of these parameters after spinal reconstructive surgery is correlated with good clinical outcome.

Maintenance of the ideal sagittal alignment allows an individual to maintain an erect posture with minimal energy expenditure. When there is progressive loss of lumbar lordosis, compensatory mechanisms involving the pelvis, hips and knees occur to extend adjacent segments of the kyphotic spine to allow for compensation of anterior translation of the axis of gravity. However, this compensatory mechanism may potentially result in adverse effect. One of the main disabilities in ASD patients with sagittal imbalance is their decreased walking tolerance. The change in the spinal alignment along with these compensatory mechanisms may result in an inefficient gait worsening their walking tolerance.

Few studies in the literature have investigated the changes in gait pattern in patients with sagittal imbalance. Of those, the patient group was heterogeneous, and the only criterion of sagittal imbalance was a positive sagittal vertical axis (SVA), which the investigators now know is not a complete assessment of the sagittal alignment. The investigators propose to study the change in gait pattern in individuals with abnormal spinopelvic parameters, and how this may affect their quality of lives.

ELIGIBILITY:
Inclusion Criteria:

All patients diagnosed with ASD, fulfilling the following radiographic criteria based on whole spine lateral film are eligible for recruitment:

* SVA bigger than 47mm
* Pelvic tilt (PT) bigger than 22deg
* Pelvic incidence (PI) - lumbar lordosis (LL) bigger than 11deg

Exclusion Criteria:

* If the aetiology of the ASD of the patient is neuromuscular origin
* other pathologies that may affect their gait such as previous trauma or surgeries to the pelvis or the lower limbs and joint replacements
* inability to walk without aids for short distances

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diagnosis of ADS will be recruited in this study conducted by the Department of Orthopaedics and Traumatology.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of sagittal imbalance on the gait cycle using reflective surface markers | 1 year
  To evaluate the effect of sagittal imbalance on the gait cycle using reflective surface markers

SECONDARY OUTCOMES:
Investigate the difference in gait kinematics between normal and abnormal sagittal balance using reflective surface markers | 1 year
  To investigate the difference in gait kinematics between normal and abnormal sagittal balance using reflective surface markers
Investigate the efficiency in gait differences between normal and abnormal sagittal balance using reflective surface markers | 1 year
  To investigate the efficiency in gait differences between normal and abnormal sagittal balance using reflective surface markers
Investigate different muscle recruitment in gait cycles between normal and abnormal sagittal balance using a submaximal graded exercise test | 1 year
  To investigate different muscle recruitment in gait cycles between normal and abnormal sagittal balance using a submaximal graded exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kenny Kwan, BMBCh(Oxon), Principal Investigator — The University of Hong Kong
Locations (1):
- Duchess of Kent Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho KJ, Suk SI, Park SR, Kim JH, Kang SB, Kim HS, Oh SJ. Risk factors of sagittal decompensation after long posterior instrumentation and fusion for degenerative lumbar scoliosis. Spine (Phila Pa 1976). 2010 Aug 1;35(17):1595-601. doi: 10.1097/BRS.0b013e3181bdad89. PMID 20386505
- [Background] Glassman SD, Berven S, Bridwell K, Horton W, Dimar JR. Correlation of radiographic parameters and clinical symptoms in adult scoliosis. Spine (Phila Pa 1976). 2005 Mar 15;30(6):682-8. doi: 10.1097/01.brs.0000155425.04536.f7. PMID 15770185
- [Background] Glassman SD, Bridwell K, Dimar JR, Horton W, Berven S, Schwab F. The impact of positive sagittal balance in adult spinal deformity. Spine (Phila Pa 1976). 2005 Sep 15;30(18):2024-9. doi: 10.1097/01.brs.0000179086.30449.96. PMID 16166889
- [Background] Smith JS, Bess S, Shaffrey CI, Burton DC, Hart RA, Hostin R, Klineberg E; International Spine Study Group. Dynamic changes of the pelvis and spine are key to predicting postoperative sagittal alignment after pedicle subtraction osteotomy: a critical analysis of preoperative planning techniques. Spine (Phila Pa 1976). 2012 May 1;37(10):845-53. doi: 10.1097/BRS.0b013e31823b0892. PMID 22024904
- [Background] Le Huec JC, Faundez A, Dominguez D, Hoffmeyer P, Aunoble S. Evidence showing the relationship between sagittal balance and clinical outcomes in surgical treatment of degenerative spinal diseases: a literature review. Int Orthop. 2015 Jan;39(1):87-95. doi: 10.1007/s00264-014-2516-6. Epub 2014 Sep 6. PMID 25192690
- [Background] Barrey C, Roussouly P, Le Huec JC, D'Acunzi G, Perrin G. Compensatory mechanisms contributing to keep the sagittal balance of the spine. Eur Spine J. 2013 Nov;22 Suppl 6(Suppl 6):S834-41. doi: 10.1007/s00586-013-3030-z. Epub 2013 Sep 20. PMID 24052406
- [Background] Engsberg JR, Bridwell KH, Reitenbach AK, Uhrich ML, Baldus C, Blanke K, Lenke LG. Preoperative gait comparisons between adults undergoing long spinal deformity fusion surgery (thoracic to L4, L5, or sacrum) and controls. Spine (Phila Pa 1976). 2001 Sep 15;26(18):2020-8. doi: 10.1097/00007632-200109150-00016. PMID 11547203
- [Background] Sarwahi V, Boachie-Adjei O, Backus SI, Taira G. Characterization of gait function in patients with postsurgical sagittal (flatback) deformity: a prospective study of 21 patients. Spine (Phila Pa 1976). 2002 Nov 1;27(21):2328-37. doi: 10.1097/00007632-200211010-00005. PMID 12438980
- [Background] Gottipati P, Fatone S, Koski T, Sugrue PA, Ganju A. Crouch gait in persons with positive sagittal spine alignment resolves with surgery. Gait Posture. 2014;39(1):372-7. doi: 10.1016/j.gaitpost.2013.08.012. Epub 2013 Aug 18. PMID 24011797
- [Background] Romei M, Galli M, Motta F, Schwartz M, Crivellini M. Use of the normalcy index for the evaluation of gait pathology. Gait Posture. 2004 Feb;19(1):85-90. doi: 10.1016/s0966-6362(03)00017-1. PMID 14741307
- [Background] Syczewska M, Dembowska-Baginska B, Perek-Polnik M, Kalinowska M, Perek D. Gait pathology assessed with Gillette Gait Index in patients after CNS tumour treatment. Gait Posture. 2010 Jul;32(3):358-62. doi: 10.1016/j.gaitpost.2010.06.006. Epub 2010 Jul 13. PMID 20630761